CLINICAL TRIAL: NCT04898712
Title: Tranexamic Acid in the Treatment of Residual Chronic Subdural Hematoma: An Observer-blinded, Randomized Controlled Trial
Brief Title: Tranexamic Acid in the Treatment of Residual Chronic Subdural Hematoma -2
Acronym: TRACE-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-232
Record Dates: First submitted 2021-05-12; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: Tranexamic acid; Chronic Subdural Hematoma; Neurosurgery
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid Arm (Experimental): Participants in the experimental arm will receive tranexamic acid (TXA) during surgery for CSDH evacuation with a single 1000mg intraoperative intravenous (IV) dose. Participants with a body weight 60-100kg will also receive a post-operative dose regimen of 500 mg TXA orally, 3 times a day (TID).
  Weight deviations from this body weight range will be considered with a dose adjustment of 1000mg TXA two times a day (BID) for a body weight >100 kg, and 500 mg TXA BID for body weight <60kg.
  Interventions: Drug: Tranexamic Acid 500 MG
- Placebo Control Arm (Placebo Comparator): Participants in the control arm will placebo according to the same administration regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Tranexamic Acid 500mg oral tablets
  Arms: Tranexamic Acid Arm
Drug: Placebo — The placebo will consist of an identical capsule to over-encapsulated tranexamic acid oral tablet entirely filled with microcrystalline cellulose, and sealed.
  Arms: Placebo Control Arm

SUMMARY:
Chronic subdural hematoma (CSDH), a common disease after minor head trauma, is characterized by blood collection in the subdural space, which can result in severe neurological impairment. The current standard of care is the surgical evacuation of CSDH. Although clinical and surgical outcomes are satisfying in most cases, considerable morbidity, mortality and recurrence rates of 3-31% are frequently reported. Therefore a non-surgical approach to treat CSDH is desirable. Tranexamic acid (TXA), an antifibrinolytic drug, has been shown to decrease hematoma volume in a small cohort of CSDH patients. The present study is designed to test the hypothesis that TXA can reduce the volume of CSDH. Volume measurements of residual CSDH after burr-hole surgery will be performed to quantify treatment success. The trial is designed as a double-blinded randomized controlled trial, where half of the patients will be assigned to daily intake of TXA, whereas the other half will receive placebo. The primary endpoint is defined as volume change in milliliter after 4-8 weeks of treatment. Secondary endpoints are hematoma volume at 8-12 weeks, patient safety, the number of patients with resolution of the CSDH after 4-8 and 8-12 weeks of study participation, the neurological outcome, the rate of reoperation, the time to reoperation, drug safety and compatibility, and participant quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic subdural hematoma (CSDH)
* Written informed consent (patient, power of attorney or substitute decision maker)
* Competence to take study medication properly and regularly or access to caregiver that is able to comply with accurate study medication administration

Exclusion Criteria:

* Hypersensitivity to TXA or any of the ingredients
* Pregnancy
* Irregular menstrual bleeding with unidentified cause
* Acquired colour vision disturbances
* Acute and chronic renal insufficiency indicated by GFR ≤ 30 mL/min
* Hematuria, caused by diseases of renal parenchyma
* Concomitant intake of hormonal contraceptives, factor IX complex concentrates, and anti-inhibitor coagulant concentrates (factor VII, activated factor IX)
* History of angioplasty with cardiac stent placement, or cardiac (including mechanical) valve placement
* Active history of stroke (hemorrhagic and ischemic), or subarachnoid hemorrhage, within the past 6 months
* Consumption coagulopathy/disseminated intravascular coagulation (DIC) in the last 7 days
* History of malignant brain tumors (glioma, metastasis and others) or seizures within the 6 months
* Contraindication to stopping full therapeutic doses of non-ASA antiplatelets, warfarin, rivaroxaban, apixaban, dabigatran, or other anticoagulant for 2 weeks after surgery
* Inability of oral drug intake or missing support to guarantee oral drug intake
* SDH as caused by intracranial hypotension resulting from CSF shunt placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Chronic subdural hematoma volume change | At 4-8 weeks
  Change in hematoma volume in mL according to CT-scan-based volume measurements comparing hematoma on CT scan performed at 4-8 weeks to hematoma on immediate post-operative CT scan.

SECONDARY OUTCOMES:
Chronic subdural hematoma volume change | At 12 weeks
  Change in hematoma volume in mL according to CT-scan-based volume measurements comparing hematoma on CT scan performed at 4-8 weeks to hematoma on immediate post-operative CT scan.
Rate of adverse events (AEs) | At 4, 8, and 12 weeks
  Adverse events investigated include:
  * suspected stroke
  * myocardial infarction
  * deep vein thrombosis
  * thromboembolic events
  * decline in renal function
  * new-onset neurological deterioration
  Serious adverse events include:
  * evidence of stroke
  * myocardial infarction
  * deep vein thrombosis
  * thromboembolic events
  * convulsions
  * severe allergic reactions
  * evidence of retinal degeneration
  * necessity of hospital admission
  * mortality
36-Item Short Form Survey (SF-36) | At 4, 8, 12 weeks
  Questionnaire assessing patient quality of life outcome profile
National Institutes of Health Stroke Scale (NIHSS) | At 4, 8, and 12 weeks
  Change in National Institutes of Health Stroke Scale (NIHSS) score (neurological outcome) at 4-8 weeks and 8-12 weeks, compared to the baseline visit score
  Minimum scale score: 0; Maximum scale score: 42. Higher score means worse neurological impairment.
Modified Rankin Scale (mRS) | At 4, 8, and 12 weeks
  Change in Modified Rankin Scale (mRS) score (neurological outcome) at 4-8 weeks and 8-12 weeks, compared to the baseline visit score
  Minimum scale score: 0 (no symptoms); Maximum scale score: 6 (death). Higher score means worse neurological outcome.
Markwalder's grading scale (MGS) | At 4, 8, and 12 weeks
  Change in Markwalder's grading scale (MGS) score (neurological outcome) at 4-8 weeks and 8-12 weeks, compared to the baseline visit score
  Minimum scale score: 0 (normal); Maximum scale score: 4. Higher score means worse neurological outcome.
Rate of re-operation | At 4, 8, and 12 weeks
  Rate of re-operation during study course due to hematoma enlargement or other significant cause
Time to reoperation | At 4, 8, and 12 weeks
  Time to reoperation during study course due to hematoma enlargement or other significant cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Cusimano, MD, PhD, Principal Investigator — St. Michael's Hospital / University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No